CLINICAL TRIAL: NCT06667180
Title: Effects of Low-intensity Transcranial Magnetic Stimulation on Major Depressive Disorder, and on 5-hydroxyindoleacetic Acid and Brain-derived Neurotrophic Factor Levels
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Olga Estefania Escobar Florez, Principal investigator, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEPIUG-P35-2023; R-2024-785-001 (Registry Identifier: National Committee for Scientific Research)
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Depression - Major Depressive Disorder; Transcranial Magnetic Stimulation; Placebo
Keywords: accelerated low-intensity transcranial magnetic stimulation; Major depressive disorder; depression; brain-derived neurotrophic factor; 5-hydroxyindoleacetic acid
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-intensity TMS (Experimental): This group will receive the real low-intensity TMS
  Interventions: Device: Low-intensity TMS
- Sham low-intensity TMS (Placebo Comparator): This group will receive the simulation of the low-intensity TMS
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Low-intensity TMS — Low-intensity TMS will be applied for 4 days, 5 daily sessions of 200 s with 10-minute intersession intervals at a field intensity of 2-4 mT and frequency of 50 Hz in theta bursts.
  Arms: Low-intensity TMS
Device: Transcranial Magnetic Stimulation Sham — The control group will receive the simulation of low-intensity TMS without magnetic field induction.
  Arms: Sham low-intensity TMS

SUMMARY:
The goal of this randomised clinical trial is to evaluate the effects of transcranial magnetic stimulation (TMS) on major depressive disorder (MDD) and on the levels of 5-hydroxyindoleacetic acid (5-HIAA) and brain-derived neurotrophic factor (BDNF). TMS works to treat MDD by using low-intensity magnetic fields to modulate certain areas of the brain, activating them which can help improve the mood of those suffering from the disorder. Final metabolites of serotonin such as 5-HIAA and growth factors such as BDNF will also be studied before starting the intervention and at the end to check if there is a significant change in their concentration. Likewise, its safety will be evaluated by monitoring the symptoms that they present at the end of the intervention and one month later. The main questions that are intended to be answered are:

* Does low-intensity TMS reduce depressive symptoms in patients with MDD?
* Does low-intensity TMS significantly change the initial and final concentrations of 5-HIAA and BDNF?
* What adverse effects might patients who are exposed to low-intensity TMS experience? The researchers will compare low-intensity and accelerated TMS with sham TMS to see if low-intensity TMS works to treat MDD.

Participants:

* Will undergo an initial clinical assessment to confirm the disorder, comorbidities, and general health status.
* A 5 mL blood sample will be taken before starting the intervention.
* Low-intensity TMS will be applied for 4 days, 5 daily sessions of 200 s with 10-minute intersession intervals at a field intensity of 2-4 milliTesla (mT) and frequency of 50 Hz in theta bursts. Symptoms will be monitored daily.
* A 5 mL blood sample will be taken at the end of the intervention and general health status clinimetrics will be reapplied.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* Both sexes.
* Those who have a diagnosis of MDD previously made by the treating psychiatrist (considering time since diagnosis and recurrence of episodes).
* Those who continue with their respective treatment and attend follow-up consultations at the health facility.
* Those who do not have a history of epilepsy, schizophrenia, neurosurgeries.
* Those who do not have metal plates anywhere in the skull, neck, chest and shoulder.
* Those who do not use pacemakers.
* Those who do not take hormone substitutes.
* Those who agree to participate in the research.

Exclusion Criteria:

* Those who are pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-08-26 (Estimated)

PRIMARY OUTCOMES:
Improvement in symptoms of depression | From admission until the end of the 4 days of intervention and one month after the end of the intervention
  Improvement in depression symptoms, assessed by the Hamilton Depression Rating Scale (HAM-D17) which measures the severity of depression symptoms.

SECONDARY OUTCOMES:
Changes in serum concentrations of 5-HIAA and BDNF | From admission until the end of the 4 days of intervention.
  5-HIAA and BDNF are neurochemical biomarkers that may correlate with response to depression treatment.

OTHER OUTCOMES:
Subjective changes in patient health | From admission until the end of the 4 days of intervention and one month after the end of the intervention
  Evaluates the perception of patients' depressive symptoms using a self-assessment scale, complementing the primary measure
Changes in sleep quality | From admission and one month after the end of the intervention
  It assesses sleep quality and detects possible improvements in sleep as an additional effect of low-intensity TMS, its improvement may indicate a secondary benefit of the treatment.
Changes in physical activity level | From admission until the end of the 4 days of intervention and one month after the end of the intervention
  The International Physical Activity Questionnaire provides information about changes during the intervention week in the patient's physical activity intensity.
Changes in the Clinical Global Impression Scale (CGI) | From admission until the end of the 4 days of intervention.
  CGI will help measure clinical changes globally.

CONTACTS AND LOCATIONS:
Overall Officials: Ma. Eugenia Garay Sevilla, PhD in medical sciences, Study Director — Universidad de Guanajuato; José M De la Roca Chiapas, PhD in medical sciences, Study Director — Universidad de Guanajuato; Blanca O Murillo Ortíz, PhD in medical sciences, Study Director — Universidad de Guanajuato; Angélica Hernández Rayas, Physics PhD, Study Chair — Universidad de Guanajuato; Olga E Escobar Florez, Master of Medical Sciences, Principal Investigator — Universidad de Guanajuato
Locations (1):
- High Specialty Medical Unit No. 1, Bajío. Mexican Social Security Institute, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) information will not be shared to ensure the privacy and confidentiality of participants, sharing IPD could expose participants to additional risks of identification, for these reasons, and to protect the rights and confidentiality of participants, we have decided not to share IPD in this study.